CLINICAL TRIAL: NCT00049322
Title: A Phase II Study Of rhuMAb VEGF (BEVACIZUMAB) In Patients With Hepatocellular Carcinoma Receiving Chemoembolization
Brief Title: Chemoembolization and Bevacizumab in Treating Patients With Liver Cancer That Cannot Be Removed With Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000258045; UCLA-0206060 (Other: UCLA); NCI-G02-2124 (Other: NCI)
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Results first posted 2016-03-15 (Estimated); Last update posted 2020-09-01 (Actual); Status verified 2016-02

CONDITIONS: Liver Cancer
Keywords: localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; adult primary hepatocellular carcinoma
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I-bevacizumab (Experimental): Patients receive bevacizumab IV over 30-90 minutes once every 2 weeks beginning 1 week prior to the first chemoembolization at a dose of 10 mg/kg. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: bevacizumab
- Arm II-chemoembolization (No Intervention): chemoembolization as part of standard of care

INTERVENTIONS:
Biological: bevacizumab — Given IV, 10mg/kg evey two weeks starting 1 week prior to the first chemoembolization.
  Patients crossed over to the Bevacizumab arm will receive Bevacizumab after week 14 at the same dose.
  Other Names: Avastin
  Arms: Arm I-bevacizumab

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as liposomal doxorubicin, cisplatin, and mitomycin, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping the cells from dividing. Chemoembolization kills tumor cells by blocking the blood flow to the tumor and keeping chemotherapy drugs near the tumor. Monoclonal antibodies, such as bevacizumab, can kill any tumor cells that are left after chemoembolization by blocking their ability to grow and spread.

PURPOSE: This randomized phase II trial is studying to see if chemoembolization followed by bevacizumab works better than chemoembolization alone in treating patients who have liver cancer that cannot be removed with surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare neovessel formation at 8 and 14 weeks after hepatic arterial chemoembolization in patients with unresectable hepatocellular carcinoma treated with bevacizumab versus no bevacizumab (observation after chemoembolization only).
* Compare time to progression, objective response rate, and tumor marker progression in patients treated with these regimens.
* Determine the pharmacokinetics of bevacizumab in patients with liver function impairment.
* Determine the toxic effects of this drug in these patients.
* Compare the cancer biomarker pattern of peripheral blood cells and plasma before and after chemoembolization in patients treated with these regimens.

OUTLINE: This is a randomized, open-label study.

All patients receive hepatic artery chemotherapy (chemoembolization) comprising doxorubicin HCl liposome, cisplatin, and mitomycin on day 8 and possibly on day 92. Patients are then randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bevacizumab IV over 30-90 minutes once every 2 weeks beginning 1 week prior to the first chemoembolization. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients do not receive bevacizumab. Patients in arm II may cross-over receive bevacizumab as in arm I if recurrent tumor is evident at week 14 by CT scan or MRI or a 50% or greater increase in AFP level has occurred since day 8 chemoembolization.

PROJECTED ACCRUAL: A total of 30 patients (15 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 year old
* Histologically or cytologically documented HCC
* Patients must have bi-dimensional measurable disease by CT or MRI scan that does not exceed 50% of the liver parenchyma
* Patients must be considered clinical candidates for chemoembolization, with at least one lesion > 3cm and no lesion > 15cm in its longest diameter
* Patients awaiting cadaveric orthotopic liver transplantation are eligible if they meet all other criteria. These patients must have a model for end-stage liver disease priority score < 28 points at entry
* Cirrhosis Child-Pugh class A or B
* Patients with documented grad III varices or prior history of UGI bleeding will require endoscopic evaluation prior to treatment under this protocol.
* Platelet count equal or greater than 60,000/μL
* Female patients must use effective contraception, be surgically sterile or be postmenopausal; male patients must be using barrier contraception or be surgically sterile
* Patients must be willing and able to comply with all study requirements and have signed the informed consent

Exclusion Criteria:

* Previous history of liver transplantation
* Fibrolamellar histology
* Prior antiangiogenesis therapy
* Presence of extrahepatic disease
* Presence of biliary obstruction defined as biliary dilatation and total bilirubin > 2.5mg/dl
* Thrombosis of the main portal vein
* Absolute contraindications to doxorubicin, mitomycin-C, cisplatin, iodinated contrast material, Avitene or dexamethasone treatment
* Other active malignancies during the past year (except for non-melanoma skin cancer or in situ carcinomas)
* ECOG PS> 2 or life expectancy < 12 weeks
* History or evidence upon physical examination of CNS disease
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, or anticipation of need for major surgical procedure within 3 months of study entry; fine needle aspirations within 7 days prior to Day 0
* Current or recent (within the 10 days prior to Day 0) use of full-dose oral or parenteral anticoagulants (except as required to maintain patency of preexisting, permanent indwelling IV catheters) or thrombolytic agent (for subjects receiving warfarin, international normalized ration of < 1.5)
* Chronic, daily treatment with aspirin (> 325mg/day) or nonsteroidal anti-inflammatory medications
* Positive pregnancy test or lactation
* Proteinuria at baseline or clinically significant impairment of renal function. Subjects unexpectedly discovered to have > 1+ proteinuria at baseline should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate < 500 mg of protein/24 hr to allow participation in the study
* Serious, nonhealing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Current or recent (within the 28 days prior to Day 0) participation in another experimental drug study
* Clinically significant cardiovascular disease, New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 1 year prior to Day 0
* Prior history of hypertensive crisis of hypertensive encephalopathy
* History of abdominal fistula or gastrointestinal perforation within 6 months prior to Day 1
* History of hemoptysis within 1 month prior to Day 1
* Significant vascular disease within 6 months prior to Day 1
* Screening clinical laboratory values:

  * ANC of < 1500/μL
  * INR of > 1.5
  * Total bilirubin of > 2.5mg/dL
  * AST or ALT > 5 times upper limit of normal
  * Serum creatinine of > 2.0 mg/dL or creatinine clearance < 45 mL/min
  * Hemoglobin of < 8.5 gm/dL
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the subject at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Britten, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Britten CD, Gomes AS, Wainberg ZA, Elashoff D, Amado R, Xin Y, Busuttil RW, Slamon DJ, Finn RS. Transarterial chemoembolization plus or minus intravenous bevacizumab in the treatment of hepatocellular cancer: a pilot study. BMC Cancer. 2012 Jan 14;12:16. doi: 10.1186/1471-2407-12-16. PMID 22244160

RESULTS

PARTICIPANT FLOW:
Recruitment Details: date of recruitment period August 2003- October 2008. Types of location: Academic medical clinics and community medical clinics.
Groups:
- Arm I (TACE-BEV Arm): Patients receive bevacizumab IV over 30-90 minutes once every 2 weeks beginning 1 week prior to the first (transarterial chemoembolization TACE)chemoembolization at a dose of 10 mg/kg. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  bevacizumab : Given IV, 10mg/kg evey two weeks starting 1 week prior to the first chemoembolization.
  Patients crossed over to the Bevacizumab arm will receive Bevacizumab after week 14 at the same dose.
- Arm II (TACE-O Arm ): Observation
Period: Overall Study
Arm/Group | Arm I (TACE-BEV Arm) | Arm II (TACE-O Arm )
Started | 15 | 15
Completed | 14 | 9
Not Completed | 1 | 6
Not completed — disease burden | 0 | 3
Not completed — Adverse Event | 1 | 0
Not completed — refused angio | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (TACE-BEV Arm) | Arm II (TACE-O Arm ) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Customized [Median (Full Range); unit: years]
  Median age | 61 [50 to 79] | 58 [49 to 75] | 59.5 [49 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Neovessel Formation as Measured by Angiogram at 14 Weeks
Description: Angiograms were assessed for changes in vascularity. The numbers indicate how many subjects in each group showed neovessel formation.
Time Frame: 14 weeks
Measure: Number; unit: participants
Arm/Group | Arm I (TACE-BEV Arm) | Arm II (TACE-O Arm )
Number analyzed (Participants) | 14 | 9
participants | 2 | 3

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) at 16 weeks (end of the core phase).
Time Frame: 16 weeks
Population: Arm I: Patients receive bevacizumab Arm II. Patients do not receive bevacizumab.
Measure: Number; unit: probablility of pfs at 16 weeks
Arm/Group | Arm I (TACE-BEV Arm) | Arm II (TACE-O Arm )
Number analyzed (Participants) | 15 | 15
probablility of pfs at 16 weeks | .79 | .19

3. Secondary Outcome: Assess the Toxicities of Bevacizumab in Patients With Liver Function Impairment
Time Frame: 16 weeks
Population: subjects that completed all 16 weeks.
Measure: Number; unit: participants
Groups:
- Arm I-bevacizumab: Patients receive bevacizumab IV over 30-90 minutes once every 2 weeks beginning 1 week prior to the first chemoembolization at a dose of 10 mg/kg. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  bevacizumab: Given IV, 10mg/kg evey two weeks starting 1 week prior to the first chemoembolization.
  Patients crossed over to the Bevacizumab arm will receive Bevacizumab after week 14 at the same dose.
Arm/Group | Arm I-bevacizumab | Arm II-chemoembolization
Number analyzed (Participants) | 15 | 14
participants
  Anemia | 3 | 6
  Anorexia | 5 | 4
  Bleeding | 8 | 1
  Constipation | 4 | 3
  Electrolyte abnormalities | 9 | 9
  Elevated alkaline phosphatase | 4 | 3
  elevated transaminases | 15 | 14
  fatigue | 9 | 8
  hyperbilirubinemia | 8 | 7
  hypertension | 6 | 4
  hypoalbuminemia | 5 | 7
  nausea and or vomiting | 6 | 9
  pain | 11 | 13
  proteinuria | 8 | 1
  pyrexia | 8 | 7
  thrombocytopenia | 7 | 10

4. Secondary Outcome: Assess Pharmakokinetics of Bevacizumab in Liver Disease
Description: bevacizumab serum concentrations
Time Frame: day 85
Measure: Mean (95% Confidence Interval); unit: micrograms/mL
Arm/Group | Arm I (TACE-BEV Arm)
Number analyzed (Participants) | 15
micrograms/mL
  Peak Day 1 | 203 [181 to 225]
  Peak Day 15 | 237 [211 to 263]
  Trough Day 15 | 35.4 [31.5 to 39.4]
  Peak Day 29 | 297 [268 to 325]
  Trough Day 29 | 74.3 [66.7 to 82]
  Peak Day 43 | 280 [232 to 328]
  Trough Day 43 | 84.7 [60.4 to 109]
  Peak Day 57 | 272 [231 to 313]
  Trough Day 57 | 97.7 [71.3 to 124]
  Peak Day 85 | 333 [300 to 366]
  Trough Day 85 | 119 [95.4 to 142]
  Day 8 | 83.2 [71.7 to 94.6]
  Day 11 | 60.9 [53.2 to 68.6]

5. Secondary Outcome: Measure (Vascular Endothelial Growth Factor)VEGF Before and After TACE With and Without Bevacizumab
Time Frame: 21 days after TACE
Measure: Number; unit: fold change
Arm/Group | Arm I (TACE-BEV Arm)
Number analyzed (Participants) | 15
fold change
  1 hour | .053
  24 hours | .167
  48 hours | .161
  72 hours | .048
  360 hours | .039
  528 hours | .063
  696 hours | .06

ADVERSE EVENTS:
Groups:
- Arm I: Patients receive bevacizumab IV over 30-90 minutes once every 2 weeks beginning 1 week prior to the first chemoembolization at a dose of 10 mg/kg. Courses repeat every 2 weeks in the absence of disease progression or unacceptable toxicity.
  bevacizumab: Given IV, 10mg/kg evey two weeks starting 1 week prior to the first chemoembolization.
  Patients crossed over to the Bevacizumab arm will receive Bevacizumab after week 14 at the same dose.
- Arm II: Patients do not receive bevacizumab
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 5/15 | 1/14
Other Adverse Events (participants affected / at risk) | 15/15 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=15) | Arm II (N=14)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0) — probable variceal bleed
Hematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Gastric Ulcers, Confusion
Partial Small Bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Liver Failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
altered mental status (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=15) | Arm II (N=14)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 6 (6)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Bleeding (Vascular disorders) | 8 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4) | 3 (3)
Electrolyte Abnormalities (Metabolism and nutrition disorders) | 9 (9) | 9 (9)
Elevated Alkaline Phosphatase (Hepatobiliary disorders) | 4 (4) | 3 (3)
Elevated Transaminases (Hepatobiliary disorders) | 15 (15) | 14 (14)
Fatigue (General disorders) | 9 (9) | 8 (8)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 8 (8) | 7 (7)
Hypertension (Cardiac disorders) | 6 (6) | 4 (4)
Hypoalbuminemia (Blood and lymphatic system disorders) | 5 (5) | 7 (7)
Nausea and or Vomiting (Gastrointestinal disorders) | 6 (6) | 9 (9)
Pain (General disorders) | 11 (11) | 13 (13)
Proteinuria (Renal and urinary disorders) | 8 (8) | 1 (1)
Pyrexia (General disorders) | 8 (8) | 7 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (7) | 10 (10)

LIMITATIONS AND CAVEATS:
Size of study limits any strong conclusions regarding efficacy.Since this study was first designed and implemented, there have been many advances in the field, including confirmation of proof of principal for anti-angiogenic agents in advanced HCC.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No